CLINICAL TRIAL: NCT02528162
Title: Evaluation of Knowledge Regarding Gestational Diabetes and Evaluation of (Group) Education for Gestational Diabetes
Brief Title: Evaluation of Education for Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: the ELENA study
Record Dates: First submitted 2015-08-06; First posted 2015-08-19 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2017-11

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; education
MeSH Terms: conditions — Diabetes, Gestational | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: education — Evaluation of education for GDM

SUMMARY:
Prospective observational cohort study of women with gestational diabetes (GDM) based on the 'International Association of Pregnancy Study Groups' (IADPSG) criteria. The overall aim is to evaluate the knowledge regarding GDM of women with GDM and to evaluate the satisfaction of women with GDM about the education they receive (given in group or individually). Normal routine care is followed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years diagnosed with GDM in the university hospital Leuven.

Exclusion Criteria:

* Women who received bariatric surgery.
* Women with pregestational diabetes or diagnosed with diabetes during early pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women diagnosed with GDM based on the IADPSG criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the knowledge regarding GDM with a self-designed questionnaire | over a 2-4 week period
Scale (0 to 3) with questionnaire on depression (CES-D ) | over a 2-4 week period
Evaluation of satisfaction with education and Diabetes Treatment Satisfaction Questionnaire | over a 2-4 week period
Scale (1-4) with questionnaire on anxiety (six-item short form STAI) | over a 2-4 week period

SECONDARY OUTCOMES:
The prevalence of GDM based on the IADPSG criteria | at 24-28 weeks of pregnancy
Composite endpoint of glycaemic control, weight, gestational weight gain and pregnancy outcomes | over a period of 16 weeks
The frequency of insulin therapy for GDM | over a period of 16 weeks
The time between the glucose challenge test and oral glucose tolerance test | at 24-28 weeks of pregnancy
The frequency of an HbA1c ≥6.5% | at 24-28 weeks of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium